CLINICAL TRIAL: NCT02540759
Title: Study of the Effect of Dose of Buglossoides Arvensis Oil on Eicosapentaenoic Acid Accrual and on the Inflammatory Response
Brief Title: Effect of Dose of Buglossoides Oil on EPA Accrual and on the Inflammatory Response
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Réseau de Santé Vitalité Health Network (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: HC-NNHPD-213421
Record Dates: First submitted 2015-08-24; First posted 2015-09-04 (Estimated); Last update posted 2016-03-11 (Estimated); Status verified 2016-03

CONDITIONS: Healthy
Keywords: Buglossoides arvensis; vegetable oil; omega-3 fatty acids; participants

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- High oleic sunflower oil (HOSO) (Placebo Comparator): 10 ml HOSO/day in a single dose, 28 days
  Interventions: Dietary Supplement: High Oleic Sunflower Oil
- High dose Buglossoides oil (Experimental): 10 ml Buglossoides oil/day in a single dose, 28 days
  Interventions: Dietary Supplement: Buglossoides oil
- Medium dose Buglossoides oil (Experimental): 6 ml Buglossoides oil + 4 ml HOSO/day in a single dose, 28 days
  Interventions: Dietary Supplement: Buglossoides oil; Dietary Supplement: High Oleic Sunflower Oil
- Low dose Buglossoides oil (Experimental): 3 ml Buglossoides oil + 7 ml HOSO/day in a single dose, 28 days
  Interventions: Dietary Supplement: Buglossoides oil; Dietary Supplement: High Oleic Sunflower Oil

INTERVENTIONS:
Dietary Supplement: Buglossoides oil
  Other Names: Ahiflower
  Arms: High dose Buglossoides oil; Low dose Buglossoides oil; Medium dose Buglossoides oil
Dietary Supplement: High Oleic Sunflower Oil
  Other Names: HOSO
  Arms: High oleic sunflower oil (HOSO); Low dose Buglossoides oil; Medium dose Buglossoides oil

SUMMARY:
The effect of various doses of Buglossoides oil on the accrual of eicosapentaenoic acid (EPA) in blood and circulating cells will be investigated.

ELIGIBILITY:
Inclusion Criteria:

1. Men or non-pregnant women, using an effective form of birth control (such as oral contraceptives, injectable contraceptives or the barrier method such as a intrauterine device (IUD) with a spermicide, a diaphragm with a spermicide, a condom with a spermicide or a sponge with a spermicide) for at least 3 months prior to entry into the study and continuing during participation in the study.
2. 18 to 65 years of age, inclusive.
3. Body mass index (BMI) 18 - 39.9 kg/m2
4. Subject is willing to avoid alcohol consumption for 24h prior to every clinic visit.
5. The subject will not modify smoking habits during supplementation period.
6. No significant medical conditions that in the opinion of the qualified physician, would preclude the subject's participation in the study.
7. Signed informed consent.
8. Willing to follow all study procedures including study visits, fasting blood draws, stable body weight, normal eating habits, current activity level, and compliance with study preparation.
9. Willing to not consume fish, crustaceans and shellfish for the duration of the study.

Exclusion Criteria:

1. Pregnancy or lactation. Women trying to conceive. Women who will try to conceive who are unwilling to commit to the use of a medically approved form of contraception throughout the study period. Method of contraception must be recorded in the case report file.
2. Individual has a condition the study physician believes would interfere with the participant's ability to provide informed consent, comply with his responsibilities during the study, which might confound the interpretation of the study results or put the person at undue risk.
3. Medical conditions including an active peptic ulcer, inflammatory bowel disease, or gastrointestinal bleeding and any medical condition or prior gastrointestinal surgery that could influence absorption, metabolism or excretion of the study supplement.
4. History or presence of significant, renal, hepatic, gastrointestinal, pulmonary, biliary, neurological or endocrine disorders.
5. History or presence of cancer in the past 2 yrs, except for non-melanoma skin cancers (e.g. basal or squamous cell carcinoma of the skin).
6. Clinically significant abnormal laboratory test results including but not limited to LDL-cholesterol ≥ 4.1mM, triglyceride levels ≥3.95mM, fasting creatinine ≥ 1.5 mg/dL, alanine transaminase or aspartate aminotransferase ≥ 1.5X the upper limit of normal.
7. Currently being treated for angina, arrhythmia and/or congestive heart failure. History of myocardial infarction or stroke.
8. Uncontrolled hypertension (resting systolic blood pressure ≥ 160 mmHg or diastolic blood pressure ≥ 100 mmHg).
9. Type 1 or 2 diabetes. Fasting glucose ≥ 100 mg/dL. HbA1c ≥ 6.0.
10. If a smoker, subject smokes no more than 1 pack (20 cigarettes) daily.
11. History (within 12 months) or current alcohol or substance abuse (no more than 14 consumptions per week; 1 consumption= 12 oz beer, 5 oz wine, 1.5 oz distilled spirits).
12. Use of any lipid-altering medications (statins, bile acid sequestrants, cholesterol absorption inhibitors, fibrates, over the counter and prescription formulations of niacin).
13. Unstable use of thyroid medication. Stable, treated hypothyroidism is not an exclusion criteria.
14. Use of any weight loss or lipid metabolism medication/supplement/program (including lipase inhibitors) within 1 month of study period OR weight gain or loss > 2 kg in the past 3 months.
15. Currently taking fish oil or any other omega-3 or omega-6 polyunsaturated fatty acids (PUFA) supplement/drug within one month of Visit 1 and throughout the study. Consumption of fatty fish (salmon, herring, mackerel, albacore tuna, and sardines) more than 2X a month within one month of visit 1 and throughout the study period. Consumption (more than twice a month) of any EPA/DHA enriched foods (e.g. docosahexaenoic acid (DHA)-enriched eggs) within one month of Visit 1. Unwillingness to avoid all fish including shellfish and crustaceans throughout the study period.
16. Use of alpha-linolenic acid-containing seeds and oils such as flax seed, chia seed, perilla seed, hemp, spirulina, walnut, mustard seed or black currant seeds/oil within one month of Visit 1 and throughout the study.
17. Use of an investigational product within the previous 30 days.
18. Has donated blood up to 4 weeks before the start of the study. Not willing to cease being a blood donor during the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2015-09; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Plasma eicosapentaenoic concentration (EPA) | Day 28
  Expressed as μmol/L plasma

SECONDARY OUTCOMES:
Plasma 20:4n-3 | Day 28
  Expressed as μmol/L plasma
Plasma docosapentaenoic acid (DPA) | Day 28
  Expressed as μmol/L plasma
Plasma 20:4n-3, EPA and DPA individually as % of total fatty acids | Day 28
Mononuclear cell 20:4n-3, EPA and DPA individually as % of total fatty acids | Day 28
Fasting serum chemistry: glucose | Day 28
Fasting serum chemistry: calcium | Day 28
Fasting serum chemistry: sodium | Day 28
Fasting serum chemistry: potassium | Day 28
Fasting serum chemistry: blood urea nitrogen | Day 28
Fasting serum chemistry: creatinine | Day 28
Fasting serum chemistry: alkaline phosphatase | Day 28
Fasting serum chemistry: aspartate aminotransferase | Day 28
Fasting serum chemistry: gamma-glutamyltransferase | Day 28
Fasting serum chemistry: total bilirubin | Day 28
Fasting serum chemistry: amylase | Day 28
Fasting serum chemistry: uric acid | Day 28
Fasting serum chemistry: albumin | Day 28
Fasting hematology: white blood cell count | Day 28
Fasting hematology: neutrophil count | Day 28
Fasting hematology: red blood cell count | Day 28
Fasting hematology:hemoglobin | Day 28
Fasting hematology: hematocrit | Day 28
Fasting hematology: platelet count | Day 28
Fasting blood lipid profile: triglycerides | Day 28
Fasting blood lipid profile: total cholesterol | Day 28
Fasting blood lipid profile: low density lipoprotein cholesterol (LDL-c) | Day 28
Fasting blood lipid profile: non-high density lipoprotein-cholesterol (non-HDL-c) | Day 28
Fasting blood lipid profile: HDL-c | Day 28
Fasting serum chemistry: chloride | Day 28
Estimated glomerular filtration rate | Day 28
Fasting hematology profile: mean corpuscular volume | Day 28
Fasting hematology profile: mean corpuscular hemoglobin | Day 28
Fasting hematology profile: mean corpuscular hemoglobin concentration | Day 28
Fasting hematology profile: red cell distribution width | Day 28
Fasting hematology profile: mean platelet volume | Day 28
Fasting hematology profile: lymphocyte concentration | Day 28
Fasting hematology profile: monocyte count | Day 28
Fasting hematology profile: eosinophil count | Day 28
Fasting hematology profile: basophil count | Day 28
Fasting hematology profile: Immature granulocytes count | Day 28
Fasting hematology profile: immature granulocytes (% white blood cell (WBC)) | Day 28
Fasting hematology profile: neutrophil (% WBC) | Day 28
Fasting hematology profile: lymphocyte (% WBC) | Day 28
Fasting hematology profile: monocytes (% WBC) | Day 28
Fasting hematology profile: eosinophil (% WBC) | Day 28
Fasting hematology profile: basophil (% WBC) | Day 28
Urinalysis: appearance | Day 28
Urinalysis: density | Day 28
Urinalysis: leukocyte esterase | Day 28
Urinalysis: nitrites | Day 28
Urinalysis: pH | Day 28
Urinalysis: protein | Day 28
Urinalysis: glucose | Day 28
Urinalysis: acetone | Day 28
Urinalysis: blood | Day 28
Urinalysis: urobilinogen | Day 28

OTHER OUTCOMES:
Cytokine production following ex vivo stimulation: interferon-gamma | Day 28
Cytokine production following ex vivo stimulation: interleukin-1beta | Day 28
Cytokine production following ex vivo stimulation: interleukin-6 | Day 28
Cytokine production following ex vivo stimulation: interleukin-8 | Day 28
Cytokine production following ex vivo stimulation: interleukin-10 | Day 28
Cytokine production following ex vivo stimulation: interleukin-17A | Day 28
Cytokine production following ex vivo stimulation: interleukin-23 | Day 28
Cytokine production following ex vivo stimulation: monocyte chemoattractant protein-1 | Day 28
Cytokine production following ex vivo stimulation: tumor necrosis factor-alpha | Day 28

CONTACTS AND LOCATIONS:
Overall Officials: Marc Surette, PhD, Principal Investigator — Université de Moncton, Moncton, NB, Canada
Locations (1):
- Université de Moncton, Moncton, New Brunswick, Canada